CLINICAL TRIAL: NCT06143956
Title: A Master Protocol for a Randomized, Controlled, Clinical Trial of Multiple Interventions for Chronic Weight Management in Adult Participants With Obesity or Overweight
Brief Title: A Master Protocol Study (LY900038) of Multiple Intervention-Specific-Appendices (ISAs) in Adult Participants With Obesity or Overweight
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 18685; W8M-MC-CWMM (Other: Eli Lilly and Company); W8M-MC-OXA1 (Other: Eli Lilly and Company); W8M-MC-LAA1 (Other: Eli Lilly and Company); W8M-MC-LAA2 (Other: Eli Lilly and Company); W8M-MC-GN01 (Other: Eli Lilly and Company); W8M-MC-GN02 (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-11-06; First posted 2023-11-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — mazdutide; Tirzepatide

STUDY DESIGN:
Intervention Model Description: The CWMM protocol includes screening assessments plus a framework for the subsequent intervention, which is the primary purpose of the protocol.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- LY3305677 Obesity ISA OXA1 (Experimental): Participants will receive LY3305677 or placebo subcutaneously (SC).
  Each ISA will detail the intervention specific analysis.
  Interventions: Drug: LY3305677; Drug: Placebo
- LY3841136 Obesity ISA LAA1 (Experimental): Participants will receive LY3841136 or placebo SC.
  Each ISA will detail the intervention specific analysis.
  Interventions: Drug: LY3841136; Drug: Placebo
- LY3841136 Obesity ISA LAA2 (Experimental): Participants will receive LY3841136, tirzepatide and placebo SC.
  Each ISA will detail the intervention specific analysis.
  Interventions: Drug: LY3841136; Drug: Tirzepatide; Drug: Placebo
- LY3549492 Obesity ISA GN01 (Experimental): Participants will receive LY3549492 orally.
  Each ISA will detail the intervention specific analysis.
  Interventions: Drug: Placebo; Drug: LY3549492
- LY3549492 Obesity ISA GN02 (Experimental): Participants will receive LY3549492 or placebo orally.
  Each ISA will detail the intervention specific analysis.
  Interventions: Drug: Placebo; Drug: LY3549492

INTERVENTIONS:
Drug: LY3305677 — Administered SC. ISA specific interventions will be listed in the ISA.
  Arms: LY3305677 Obesity ISA OXA1
Drug: LY3841136 — Administered SC. ISA specific interventions will be listed in the ISA.
  Arms: LY3841136 Obesity ISA LAA1; LY3841136 Obesity ISA LAA2
Drug: Tirzepatide — Administered SC. ISA specific interventions will be listed in the ISA.
  Arms: LY3841136 Obesity ISA LAA2
Drug: Placebo — Administered SC. ISA specific interventions will be listed in the ISA.
Drug: LY3549492 — Administered orally. ISA specific interventions will be listed in the ISA.
  Arms: LY3549492 Obesity ISA GN01; LY3549492 Obesity ISA GN02

SUMMARY:
The purpose of this Phase-2 chronic weight management master protocol (CWMM) is to create a framework to evaluate the safety and efficacy of various investigational interventions for chronic weight management with intervention-specific appendices (ISAs). The CWMM establishes entry criteria for newly enrolled participants across the master and the ISAs. The ISAs may start independently of other ISAs as interventions become available for clinical testing. The results for the CWMM screening record will be reported when all the ISA's complete.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI)

  * ≥30 kilogram/square meter (kg/m²), or
  * ≥27 kg/m² and <30 kg/m², or with at least 1 weight-related comorbidity
* Have had a stable body weight for the 3 months prior to randomization (<5%) body weight gain and/or loss.

Exclusion Criteria:

* Have a prior or planned surgical treatment for obesity, except prior liposuction or abdominoplasty, if performed >1 year prior to screening.
* Have type 1 diabetes mellitus, latent autoimmune diabetes in adults, or history of ketoacidosis or hyperosmolar coma.
* Have poorly controlled hypertension.
* Have signs and symptoms of any liver disease other than nonalcoholic fatty liver disease.
* Have any of the following cardiovascular conditions within 3 months prior to screening:

  * acute myocardial infarction
  * cerebrovascular accident (stroke)
  * unstable angina, or
  * hospitalization due to congestive heart failure.
* Have a history of symptomatic gallbladder disease within the past 2 years.
* Have a lifetime history of suicide attempts.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1217 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Allocated to Each ISA | Baseline to Week 6
  Each ISA will detail the intervention specific analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (53):
- United States (49):
  - The Institute for Liver Health II dba Arizona Clinical Trials - Mesa, Chandler, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - Headlands Research - Scottsdale, Scottsdale, Arizona
  - The Institute for Liver Health II dba Arizona Liver Health-Tucson, Tucson, Arizona
  - NorCal Medical Research, Inc, Greenbrae, California
  - Velocity Clinical Research, Huntington Park, Huntington Park, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Northeast Research Institute (NERI), Fleming Island, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - New Horizon Research Center, Miami, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Charter Research - Winter Park, Orlando, Florida
  - Charter Research - Lady Lake, The Villages, Florida
  - Pacific Diabetes & Endocrine Center, Honolulu, Hawaii
  - Medical Research Partners, Ammon, Idaho
  - Great Lakes Clinical Trials - Ravenswood, Chicago, Illinois
  - NorthShore University Health System, Skokie, Illinois
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Cotton O'Neil Diabetes & Endocrinology, Topeka, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Knownwell, Needham, Massachusetts
  - Lucida Clinical Trials, New Bedford, Massachusetts
  - Headlands Research - Detroit, Southfield, Michigan
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Clinvest Headlands Llc, Springfield, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Dent Neurologic Institute, Amherst, New York
  - Velocity Clinical Research, Syracuse, East Syracuse, New York
  - North Suffolk Neurology, Port Jefferson Station, New York
  - Rochester Clinical Research, LLC, Rochester, New York
  - Medication Management, Greensboro, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - Lucas Research, Inc, Morehead City, North Carolina
  - Lucas Research, Inc., New Bern, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - Quality Medical Research, Nashville, Tennessee
  - IMA Clinical Research Austin, Austin, Texas
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Tekton Research - Fredericksburg Road, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Texas Valley Clinical Research, Weslaco, Texas
  - Sovah Clinical Research-River District, Danville, Virginia
  - Central Washington Health Services Association d/b/a Confluence Health, Wenatchee, Washington
- Argentina (4):
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
  - Centro Médico Viamonte, Buenos Aires
  - Consultorio de Investigación Clínica EMO SRL, Buenos Aires
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/